CLINICAL TRIAL: NCT07080190
Title: Assessment of the Role of Early Urine Alkalinization and N-Acetylcysteine Administration in the Management of Hair Dye (Paraphenylene Diamine) Intoxication
Brief Title: Early Urine Alkalinization and N-Acetylcysteine Administration in the Management of Hair Dye (Paraphenylene Diamine) Intoxication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Om koulthoum Mahmoud Abozeid Soliman, Assistant Lecturer of Forensic Medicine and Clinical Toxicology, Faculty of Medicine, South Valley University, Qena, Egypt., South Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SVU/MED/FMT010/2/22/6/412
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Urine Alkalinization; N-Acetylcysteine; Hair Dye; Paraphenylene Diamine; Intoxication

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients received early N-Acetylcysteine.
  Interventions: Drug: Early N-Acetylcysteine
- Control group (Active Comparator): Patients received late N-Acetylcysteine.
  Interventions: Drug: Late N-Acetylcysteine

INTERVENTIONS:
Drug: Early N-Acetylcysteine — Patients received N-acetyl cysteine early (at admission) in the course of treatment of acute hair dye poisoning.
  Arms: Study group
Drug: Late N-Acetylcysteine — Patients received the standard treatment of N-acetyl cysteine after starting organ affection in the course of treatment of acute hair dye poisoning.
  Arms: Control group

SUMMARY:
This study aimed to determine the role of early urine alkalinization and N-acetylcysteine administration for the prevention of renal damage following hair dye intoxication

DETAILED DESCRIPTION:
Paraphenylenediamine (PPD) is an organic compound with the formula C6H4(NH2). It is the derivative of aniline, which is a white substance that turns black on oxidation, called paraphenylaniline, which is soluble in hydrogen peroxide.

Intoxication with hair dye (PPD) has become a standard method of intentional self-harm in some parts of Africa and Asia because it is cheap and readily available in the market(5).

It can cause contact dermatitis in susceptible individuals. The glutathione (GSH) levels are depleted in PPD poisoning. The antioxidant GSH plays a vital role in the maintenance of cell viability, DNA replication, and the regulation of immune cell functions. N-acetylcysteine (NAC) acts as an antioxidant both directly as a glutathione substitute and indirectly as a precursor for glutathione.

ELIGIBILITY:
Inclusion Criteria:

* Both sexes.
* Patients presented acutely to the emergency department with an evident history and clinical features of hair dye intoxication

Exclusion Criteria:

* Renal disease.
* Hepatic disease.
* Diabetes mellitus.
* Hypertension.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Mean difference of the serum creatinine | Immediately after N-Acetylcysteine Administration (Up to 1 hour)
  Mean difference of the serum creatinine was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- South Valley university, Qina, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.